CLINICAL TRIAL: NCT06092866
Title: Digital Versus Telephone Symptom Assessment and Triage in Primary Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Veronica Milos Nymberg, Associate professor, Lund University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022-03883-01
Record Dates: First submitted 2023-08-10; First posted 2023-10-23 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Infections; Injuries; Psychiatric Disorder; Gastro-Intestinal Disorder; Skin Diseases
Keywords: triage; primary care; digital; remote; health care consumption
MeSH Terms: conditions — Infections; Wounds and Injuries; Mental Disorders; Digestive System Diseases; Skin Diseases

STUDY DESIGN:
Intervention Model Description: Randomization 1:1
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital triage (Experimental): Patients are triaged with symptom assessment by a nurse using a digital platform. They are receiving either advice for self-care, referred to other care-level or booked to a digital or physical visit on the primary health care center.
  Interventions: Behavioral: Digital triage
- Telephone triage (Active Comparator): Patients are triaged with symptom assessment by a nurse using tradition telephone. They are receiving either advice for self-care, referred to other care-level or booked to a digital or physical visit on the primary health care center.
  Interventions: Behavioral: Digital triage

INTERVENTIONS:
Behavioral: Digital triage — A registered nurse assesses the symptoms reported by the patient on the online platform and gives appropriate advice for further care using chat.
  Other Names: Symptom assessment

SUMMARY:
A 'digital-first' approach is currently under implementation in several Swedish regions.

The principles behind implementing an online service as an access way to primary care are based on an expectation that it can make access easier, direct people to appropriate levels of care, and increase both availability of heath care and cost efficiency. However, a recent Swedish report concluded that digital triage in primary care has not been investigated in a clinical real-world setting, including real patients, meaning that the benefits and risks for patients as well as on a system level remain unclear.

The aim of this trial is to study the feasibility of a larger trial that will compare digital triage and traditional telephone triage on adherence to triaged health care level, in a randomized controlled study (feasibility study, RCT). The study will recruit a total of 120 patients, of which half will be randomized to telephone triage and half to digital triage.

DETAILED DESCRIPTION:
Ten regions in Sweden are currently collaborating in the implementation of a new digital platform for digital symptom assessment and triage.

The patient's path is as following:

1. Triage to self-care. The patient will start his/her health care contact at the website www.1177.se with mobile bank identification. An algorithm-based computerized symptom checker performs the initial assessment, based on patient's self-reported complains. This initial triage can result in an auto-triage with self-care advice for non-complicated health issues.
2. Triage to digital assessment by chat with a nurse. Patients with more complex needs will be directed to the primary health care center (PHCC) where the patient is listed. There is also a central back-up unit that manages patients during out of office hours. The triage nurse can supplement the patient history with additional questions and finally determine the level of care.
3. Patients in need of further assessment are booked to a physical visit to a doctor or other health care staff, or referral to an emergency room.

Study design

Design: Feasibility study, randomized controlled study Patients: Patients referred by the online symptom checker to digital triage with a nurse and patients receiving traditional telephone triage. This study is planned to be carried out at one or more health centers where both traditional telephone triage and digital triage are used. The study will be conducted initially as a feasibility study with 30 participants in each arm and the inclusion period will continue until this number is met. A larger RCT is planned in the future, based on the feasibility study. The consent to participate will be filled in electronically by the participants in the digital triage group, and by the nurse in the telephone group (and documented in the electronic medical record).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older who is listed at the health center

Exclusion Criteria:

* Patients <18 years or parents seeking advice for their children

  * Cannot communicate in Swedish or other communication difficulties in language or writing
  * Patients without a mobile Bank identification (to log in to the platform)
  * Administrative issues, e.g. rebooking of time

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate as percentage of patients included in the study measured using data from the primary health care center | 6 months
  Percentage of patients that accept to be included in the study of all patients that contact the primary care center during the studied period of time
Drop-out rate as percentage of patients that drop-out from the trial | 6 months
  Percentage of patients that drop-out from the trial
Eligibility criteria in percentage of patients being eligible to be included in the study | 6 months
  Age 18 years or older and listed on the primary care center

SECONDARY OUTCOMES:
Adherence to recommended health care level as percentage of patients that adhere to recommended care level | 2 months
  Within 2 months after the triage contact, data collected from the regional data base
Interrater reliability | 2 months
  agreement between the care-level suggested by the online symptom checker and the care-level suggested by the nurse, data collected from the electronic medical journals

CONTACTS AND LOCATIONS:
Overall Officials: Veronica V Milos Nymberg, PhD, Principal Investigator — Lund University
Locations (1):
- Veronica Milos Nymberg, Malmo, Region Skane, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared with researchers at Lund university or other universities upon reasonable request.